CLINICAL TRIAL: NCT06569576
Title: Promoting Aging in Place Through A Wellness Program: Comparing In-person and Online Delivery
Brief Title: Promoting Aging in Place Through A Wellness Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy University (Other)
Collaborators: Yeshiva University (Other)
Responsible Party: Principal Investigator, Jeanine, Associate Professor, Mercy University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-57
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Group Meetings; Telehealth
MeSH Terms: interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: Comparing online delivery vs in-person delivery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- in-person wellness program (Experimental): The program is delivered at the senior center site.
  Interventions: Behavioral: Wellness program
- Online Wellness Program (Experimental): The program is delivered remotely. Participants join from their home environment.
  Interventions: Behavioral: Wellness program

INTERVENTIONS:
Behavioral: Wellness program — It combines seated yoga exercises, mindfulness, and social participation activities and discussions, and can be delivered in-person or via tele-health.

SUMMARY:
Study explores the impact of an eight-week Healthy Aging Wellness (HAW) group-based program delivered online and in-person to improve hope and well-being in community-dwelling older adults.

DETAILED DESCRIPTION:
Study explores the impact of an eight-week Healthy Aging Wellness (HAW) group-based program delivered online and in-person to improve hope and well-being in community-dwelling older adults. This study explores the implementation of the Healthy Aging Wellness program to support aging in place of community-dwelling older adults. It combines seated yoga exercises, mindfulness, and social activities.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* independent in everyday life
* living at home
* Mini-Mental State Examination (MMSE) > 26
* English speakers
* access to a device with a camera and reliable internet services if they were recruited for the tele-health group
* health status verified by primary care physician.

Exclusion Criteria:

* balance issues
* history of falls within the last 6 months
* medical conditions considered contra-indications to exercise
* cognitive impairments, which may make participation in the program unsafe.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-07 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Integrative Hope Scale (IHS) | up to 8 weeks
  * Self-measure of person's sense of hope
  * Scored on a scale ranging from 1 (low) to 6 (high) points
  * Total score ranges from 23 to138
Personal Wellbeing Index: 5th Edition | up to 8 weeks
  * Self-measure of person's sense of wellbeing
  * Scale from 0-10
  * higher number indicates greater satisfaction

SECONDARY OUTCOMES:
Open ended interview | up to 8 weeks
  Interviewing individuals about their experience in the program

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy University, Dobbs Ferry, New York, United States

IPD SHARING:
Plan to Share IPD: No